CLINICAL TRIAL: NCT01734551
Title: Pharmacological Treatment of Neonatal Abstinence Syndrome: Opiate Versus Non-Opiate
Brief Title: NAS Treatment - Opiate Versus Non-Opiate
Acronym: NAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henrietta Bada (Other)
Responsible Party: Sponsor-Investigator, Henrietta Bada, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0534
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Prenatal opiate exposure; neonatal withdrawal; Pharmacologic treatment
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Morphine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): Initial dose is 0.4mg/kg/day, divided every 3-4 hours, given PO with feeds. Drug is required until symptoms of withdrawal no longer cause the infant feeding, behavior, or elimination problems, up to 3 months.
  Interventions: Drug: Morphine
- Clonidine (Active Comparator): Dose is started at 5 mcg/kg/day, given PO with feeds, divided every 3-4 hours. Drug is required until symptoms of withdrawal no longer cause the infant feeding, behavior, or elimination problems, up to 3 months.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Morphine — Start at 0.4mg/kg/day (divided every 3-4 hours, given with feeds. Dose may be increased 25% of initial dose until symptoms are stable, up to 1 mg/kg/day.
  Once stable for 72 hrs, weaning may begin (decrease 10% of max dose, every other day). When total dose is <0.1mg/kg/day, may discontinue.
  Other Names: Morphine sulfate
  Arms: Morphine
Drug: Clonidine — Initial dose is 5 mcg/kg/day (divided every 3-4 hrs, given with feeds). Will increase 25% of initial dose every 12-24 hrs until stable, up to 12 mcg/kg/day. Dose is unchanged for 72 hours once stable, then may decrease by 10% every other day. If re-escalation is required, the previous dose may be used with 72 hours for stabilizing.
  Other Names: clonidine hydrochloride
  Arms: Clonidine

SUMMARY:
The purpose of this study is to compare two different medicines to treat babies with opiate withdrawal. The treatment medicines are morphine, which is an opiate, and clonidine, a non-opiate. Morphine is a narcotic medicine, with is included in most pain killers. Clonidine is another drug, but is different from morphine. It is also used for babies, and even adults for withdrawal symptoms. Both drugs are effective, but the purpose of this study is to see if one may be better than the other.

DETAILED DESCRIPTION:
Withdrawal from drugs, called Neonatal abstinence syndrome (NAS), is a group of symptoms that occurs to babies whose mother took or used drugs (prescription, addicting, illegal, pain pills, or drugs for addiction treatment) during pregnancy. Medicines the mother takes while pregnant, the baby also takes. Babies may experience withdrawal after delivery, and may need treatment. There are different ways to treat babies with withdrawal - about 50% of doctors use morphine, an opiate, to treat these babies, the rest uses other drugs, like clonidine and phenobarbitol.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Neonatal Intensive Care Unit (NICU)- Gestational age (GA) >or= 35 wks
* Known prenatal opiate exposure (maternal history, positive opiate screen, positive neonatal urine or meconium screen)
* Symptomatic with Finnegan Neonatal Abstinence Scores meeting NICU protocol for treatment

Exclusion Criteria:

* Seizures
* Major congenital malformations
* Unlikely to survive
* Parents not able to understand English

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrietta S Bada, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914
- [Derived] Bada HS, Sithisarn T, Gibson J, Garlitz K, Caldwell R, Capilouto G, Li Y, Leggas M, Breheny P. Morphine versus clonidine for neonatal abstinence syndrome. Pediatrics. 2015 Feb;135(2):e383-91. doi: 10.1542/peds.2014-2377. PMID 25624389

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine: Initial dose is 0.4mg/kg/day, divided every 3-4 hours, given PO with feeds. Drug is required until symptoms of withdrawal no longer cause the infant feeding, behavior, or elimination problems, up to 3 months.
  Morphine: Start at 0.4mg/kg/day (divided every 3-4 hours, given with feeds. Dose may be increased 25% of initial dose until symptoms are stable, up to 1 mg/kg/day.
  Once stable for 72 hrs, weaning may begin (decrease 10% of max dose, every other day). When total dose is <0.1mg/kg/day, may discontinue.
Period: Overall Study
Arm/Group | Morphine | Clonidine
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Clonidine | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Finnegan Neonatal Abstinence Scoring System
Description: Mean of total Finnegan Scores obtained every 3 hours on days 2, 7, and 14 following start of treatment; A score is a number representing the total score or sum from 21 items or symptoms or manifestations of opiate withdrawal in newborn infants. The total score ranges from 0 to 43. Reference: 1. Finnegan LP, Connaughton JF, Jr., Kron RE, et al. Neonatal abstinence syndrome: assessment and management. Addict Dis 1975;2(1-2):141-58. Although normal newborn may manifest mild symptoms that will give scores in the range of 0 to 7. A score of 8 consecutively obtained times 3 indicate that infant will benefit from treatment, in this study morphine or clonidine. A decrease in scores especially to less than 8 is suggestive of a good response to treatment.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Morphine | Clonidine
Number analyzed (Participants) | 15 | 16
scores on a scale
  Finnegan scores day 2 of treatment | 7.5 (0.35) | 8.5 (0.30)
  Finnegan scores day 7 of treatment | 6.6 (0.65) | 5.7 (0.44)
  Finnegan scores day 14 of treatment | 7.1 (1.1) | 6.7 (0.98)

2. Primary Outcome: Duration of Treatment
Description: Total number days of treatment
Time Frame: 120 days
Measure: Median (Full Range); unit: days
Arm/Group | Morphine | Clonidine
Number analyzed (Participants) | 15 | 16
days | 39 [26 to 89] | 27 [18 to 107]

3. Secondary Outcome: Neurobehavioral Performance Summary Scores From the Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS)
Description: The summary scores from the Neonatal Intensive Care Unit Network Neurobehavioral Scale (NNNS) give a measure of infant neurobehavior in the following areas (score range): habituation (1-9), regulation (2.20-7.50), attention (1.29 -8.4), Handling (0 - 1), quality of movement (1.20 - 6.20), Non-optimal reflexes (0-12), Asymmetric reflexes (0-7), arousal (2.43 - 6.67), hypertonicity (0- 8), hypotonicity (0 - 5.0), excitability (0-11), lethargy (0 - 11.0). and stress/abstinence (0. - 0.57). A higher score for each item means a higher level of the construct. For example, a higher score for hypertonicity means the infant is more hypertonic and higher score on hypotonicity means the infant is more hypotonic. No cut-off score published for normal or abnormal behavioral performance. Reference: Lester BM et al. Summary Statistics of Neonatal Intensive Care Unit Network Neurobehavioral Scale Scores From the Maternal Lifestyle Study: A Quasinormative Sample, in Pediatrics 2004; 113,668.
Time Frame: 5-10 days after treatment starts
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Morphine | Clonidine
Number analyzed (Participants) | 15 | 16
scores on a scale
  Attention | 5.06 (0.27) | 4.51 (0.26)
  Handling | 0.36 (0.06) | 0.42 (0.06)
  Quality of movement | 4.77 (0.15) | 4.92 (0.14)
  Regulation | 5.2 (0.18) | 5.26 (0.17)
  Non-optimal reflexes | 3.73 (0.42) | 4.13 (0.40)
  Asymmetric reflexes | 0.20 (0.14) | 0.00 (0.14)
  Stress/abstinence | 0.07 (0.01) | 0.08 (0.01)
  Arousal | 3.91 (0.13) | 3.95 (0.13)
  Hypertonicity | 0.40 (0.25) | 0.25 (0.24)
  Hypotonicity | 0.13 (0.13) | 0.19 (0.13)
  Excitability | 2.6 (0.53) | 2.38 (0.51)
  Lethargy | 3.6 (0.50) | 5.13 (0.03)

4. Secondary Outcome: Bayley Scales of Infant and Toddler Development Third Edition
Description: Scores obtained Bayley Scales of Infant and Toddler Development Third Edition in the developmental domains of motor, cognitive, and language. This tool for measures of motor, cognitive and language development is a series of standardized measurements and for each domain, the standardized scores have a mean of 100 and standard deviation of 15. Scores below 1 standard deviation (= or less than 84) is considered below normal. Scores above 1 standard deviation (over 115) represent higher than normal functioning in each domain The score for each domain (motor, cognitive, and language functioning) represents the full-scale score
Time Frame: 1 year of life
Population: The above number fo reach arm represents the number of subjects who came for follow-up evaluation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Morphine | Clonidine
Number analyzed (Participants) | 12 | 12
scores on a scale
  Bayley III motor | 97.6 (10.4) | 95.8 (7.2)
  Cognitive | 92.9 (8.4) | 93.3 (7.2)
  Language total | 98.0 (13.8) | 95.8 (10.4)
  Language Receptive | 101.1 (14.3) | 95.0 (12.2)
  Language Expressive | 100.0 (13.1) | 99.2 (13.6)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Daily review of inpatient care and activity. Upon discharge, electronic medical records reviewed for 3 months after infant left UK NICU. Assessments at NICU Graduate Clinic were done at 3 months
Arm/Group | Morphine | Clonidine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No